CLINICAL TRIAL: NCT00336726
Title: Neuroendocrine Dysfunction in Traumatic Brain Injury: Correlation With Cognitive Dysfunction and Repair
Status: Terminated | Type: Observational
Sponsor: Denver Research Institute (Other)
Responsible Party: Margaret Wierman, M.D., VA Medical Center
Other Study IDs: GR-735
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2004-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Traumatic Brain Injury (TBI) is a neurologic disorder cuased by physical trauma to the brain. Neuroendocrine abnormalities in these patients have been reported, including central hypogonadism within hours of the insult and eventual recovery of the hypothalamic-pituitary-gonadal axis with recovery of cognitive function to baseline. This pilot study will measure hormonal level of neuroendocine function at the time of TBI and various time points during recovery.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects having had a recent traumatic brain injury.

Exclusion Criteria:

* Currently receivng sex steroids, glucocorticoids, or have an inability to complete the neurobehavioral assessment.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male subjects having had a recent traumatic brain injury
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Wierman, MD, Principal Investigator — Dept. of Veterans Affairs/University of Colorado HSC